CLINICAL TRIAL: NCT00186446
Title: Treatment of Nicotine Dependence and Acute Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Alan Schatzberg, Professor, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GSK 103341
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Results first posted 2017-04-04 (Actual); Last update posted 2017-04-04 (Actual); Status verified 2017-02

CONDITIONS: Major Depressive Disorder; Nicotine Dependence
MeSH Terms: conditions — Depressive Disorder, Major; Tobacco Use Disorder | interventions — Bupropion

ARMS (1):
- Bupropion (Experimental)
  Interventions: Drug: bupropion and smoking cessation behavioral intervention

INTERVENTIONS:
Drug: bupropion and smoking cessation behavioral intervention

SUMMARY:
The purpose of this study is to assess the safety and feasibility of concurrent treatment of nicotine dependence (cigarette smoking) and acute depression. Participants who meet DSM-IV criteria for both nicotine dependence and acute major depression will be given pharmacological treatment for both disorders at the same time, along with a brief behavioral intervention for smoking cessation.

DETAILED DESCRIPTION:
The purpose of this study is to assess the safety and feasibility of concurrent treatment of nicotine dependence (cigarette smoking) and acute depression. Participants who meet DSM-IV criteria for both nicotine dependence and acute major depression will be given pharmacological treatment for both disorders at the same time, along with a brief behavioral intervention for smoking cessation.

ELIGIBILITY:
Inclusion Criteria:

* Age at least 18 at the beginning of the study
* Smoking at least 10 cigarettes a day (1/2 pack)
* Meets DSM-IV criteria for major depressive episode

Exclusion Criteria:

* Currently pregnant
* Currently breastfeeding
* Currently diagnosed with a seizure disorder, liver disease, kidney disease, congestive heart failure or diabetes mellitis
* History of a seizure, seizure disorder, significant head trauma or central nervous system tumor
* Family history of seizures
* Currently using intravenous drugs
* Currently using any drugs (marijuana, alcohol, cocaine, opiates, stimulants, etc.) on a daily basis
* Currently using any over-the-counter stimulants and anorectics (diet pills)
* Currently on fluoxetine (Prozac), bupropion (Wellbutrin, Wellbutrin SR, Wellbutrin XL) or any other antidepressants, monoamine oxidase inhibitors, antipsychotics, benzodiazepines, theophylline, systemic steroids or levodopa
* Currently on NRT or bupropion (Zyban)
* Current or past diagnosis of anorexia nervosa
* Previous allergic response to fluoxetine, bupropion, or NRT
* Previous failed quit attempt using NRT and bupropion in combination
* Current suicidal ideation
* Current or past psychosis, mania/hypomania, or any other Axis I or Axis II psychiatric diagnosis other than major depression and nicotine dependence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2004-06; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Lembke, MD, Study Director — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Bupropion and Smoking Cessation Behavioral Intervention: Medication for depression and behavioral intervention for smoking cessation
Period: Overall Study
Arm/Group | Bupropion and Smoking Cessation Behavioral Intervention
Started | 20
Completed | 11
Not Completed | 9

BASELINE CHARACTERISTICS:
Arm/Group | Bupropion and Smoking Cessation Behavioral Intervention
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.35 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 17
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Hamilton Depression Scale Score
Description: Utilized the Hamilton Depression Rating Scale, 21-item version to assess depressive symptoms, with a range of 0-63. Higher values indicate more depression. % Change in depression score from baseline to week 10. Negative values indicate a reduction in depression.
Time Frame: baseline to week 10
Population: 9 patients did not complete the study and we used last observation carried forward
Measure: Mean (Standard Deviation); unit: percentage of change in depression
Arm/Group | Bupropion and Smoking Cessation Behavioral Intervention
Number analyzed (Participants) | 20
percentage of change in depression | -.5322 (.27)
Statistical Analysis 1: Comparison: Bupropion and Smoking Cessation Behavioral Intervention; Test type: Superiority or Other; p < .001, t-test, 2 sided; t(19)= -8.93

2. Primary Outcome: Cessation of Smoking
Description: Carbon monoxide breath level of below 9PPM which indicates cessation of smoking.
Time Frame: Week 10
Population: Carbon monoxide levels available on 8 subjects at week 10.
Measure: Count of Participants; unit: Participants
Arm/Group | Bupropion and Smoking Cessation Behavioral Intervention
Number analyzed (Participants) | 8
Participants | 7

3. Primary Outcome: Can Depression and Smoking Cessation be Treated Simultaneously
Description: This was measured by the drop out rate during the study.
Time Frame: Dropouts over course of study
Population: Number dropped out of the study
Measure: Count of Participants; unit: Participants
Groups:
- Bupropion and Smoking Cessation Behavioral Intervention: bupropion and behavioral intervention
Arm/Group | Bupropion and Smoking Cessation Behavioral Intervention
Number analyzed (Participants) | 20
Participants | 9

ADVERSE EVENTS:
Arm/Group | Bupropion and Smoking Cessation Behavioral Intervention
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No